CLINICAL TRIAL: NCT05283629
Title: Neuroplasticity-Based Cognitive Remediation for Chemotherapy Related Cognitive Impairment Randomized Study
Brief Title: nCCR for Chemotherapy Related Cognitive Impairment Randomized Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Utah (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Vega, Primary Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211521
Record Dates: First submitted 2022-02-03; First posted 2022-03-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chemo-brain; Chemotherapy-Related Cognitive Impairment
Keywords: Chemotherapy; Cognitive Impairment; neuroplasticity-based computerized cognitive remediation; nCCR
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participants and the primary investigator are blinded to the arm of the study they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroplasticity-based Computerized Cognitive Remediation (Experimental): Behavioral: Neuroplasticity-based Computerized Cognitive Remediation Participants will engage in a computerized training program designed to support cognitive health in older adults. The program includes a variety of exercises that target basic sensory processing as well as higher-level cognitive functions. Training tasks adapt in difficulty based on individual performance and are intended to improve information processing and executive skills. Activities are delivered in a structured format and customized to participant progress.
  Interventions: Behavioral: Neuroplasticity-based Computerized Cognitive Remediation
- Active Comparison Control (Active Comparator): The active control condition is a structured, learning-based program designed to match the nCCR intervention in terms of duration, computer use, audiovisual engagement, and participant contact with research staff.
  Interventions: Behavioral: Active Control Condition

INTERVENTIONS:
Behavioral: Neuroplasticity-based Computerized Cognitive Remediation — Behavioral: Neuroplasticity-based Computerized Cognitive Remediation Participants will engage in a computerized training program designed to support cognitive health in older adults. The program includes a variety of exercises that target basic sensory processing as well as higher-level cognitive functions. Training tasks adapt in difficulty based on individual performance and are intended to improve information processing and executive skills. Activities are delivered in a structured format and customized to participant progress.
  Arms: Neuroplasticity-based Computerized Cognitive Remediation
Behavioral: Active Control Condition — The active control condition is a structured, learning-based program designed to match the nCCR intervention in terms of duration, computer use, audiovisual engagement, and participant contact with research staff.
  Arms: Active Comparison Control

SUMMARY:
The investigators propose to apply neuroplasticity-based computerized cognitive remediation (nCCR) to treat chemotherapy-related cognitive impairment (CRCI).

DETAILED DESCRIPTION:
Successes in breast cancer treatment are resulting in a growing number of cancer survivors. This has broadened the scope of care from treating the disease alone to improving the quality of life of cancer survivors. Chemotherapy-related cognitive impairment (CRCI), often referred to by patients as 'chemobrain,' is a common and highly distressful side effect of chemotherapy often reported by breast cancer survivors. Managing the symptoms of CRCI should be integrated with routine cancer care as these symptoms diminish quality of life, impair work performance, and make it more difficult for patients to follow treatment regimens. CRCI can persist for months to years following cancer treatment. However, there are currently no established treatments for CRCI.

The most commonly reported CRCI symptoms in breast cancer survivors include problems with executive functions. Executive function is a cognitive domain involved in planning, problem-solving, organization, and time management. In order to improve executive dysfunction and quality of life in breast cancer survivors, we propose to use a new brain training program called neuroplasticity-based computerized cognitive remediation (nCCR). The term 'neuroplasticity' refers to the brain's ability to modify, change, and adapt throughout life and in response to experience. Neuroplacticity can be induced through the use of focused brain training that nCCR offers. Past work demonstrates that this neuroscience-guided brain training benefits other patient populations with similar cognitive problems and has shown preliminary success in cancer survivors in a small pilot study. If successful, this treatment could have significant benefits for large numbers of breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

All participants will:

* between 35 and 80 years of age
* have been diagnosed with noninvasive or invasive breast cancer
* have undergone treatment with systemic chemotherapy within the last 1- 8 years
* endorse persistent CRCI subjective complaints
* have no active unstable medical condition
* fluent in and able to read English.

Exclusion Criteria:

Participants will be excluded for

* any active neurologic or untreated/non-remitted psychiatric disease, (e.g. active major depression or another major psychiatric disorder as described in DSM-5)
* clinically significant cognitive impairment identified on cognitive screening, diagnosis of mild cognitive impairment or dementia
* history of significant head trauma followed by persistent neurologic deficits
* history of alcohol or substance abuse or dependence within the past 2 years (DSM-5 criteria)
* any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol
* Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening
* red-green color blindness
* Use of certain CNS active medications (e.g. antidepressants) will be permitted, provided dosing has been stable for at least 3 months.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Assess whether nCCR training produces change in subjective cognitive complaints breast cancer survivors with CRCI. | 6-weeks
  Paired samples t-tests will be used to assess FACT-Cog PCI Scores. We hypothesize that nCCR treatment will improve FACT-Cog scores in breast cancer patients with persistent CRCI over 6 weeks of treatment compared to the education control group.
  The primary measure used to assess subjective cognitive performance was the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) scale and evaluates memory, concentration, mental acuity, verbal fluency, functional interference, and multitasking ability. At baseline and post-treatment visits, participants rated on a 5-point Likert scale how they assessed various aspects of their cognitive functioning over the last 7 days. Higher scores indicate better ratings of cognitive functioning. Higher scores indicate better ratings of cognitive functioning.

SECONDARY OUTCOMES:
Assess whether 6-weeks of nCCR training produces change in cognitive performance on neuropsychological measures in breast cancer survivors with CRCI. | 6-weeks
  Paired samples t-tests will be used to assess Trail Making Test performance. We hypothesize that nCCR treatment will improve Trail Making Test performance in breast cancer patients with persistent CRCI over 6 weeks of treatment compared to the education control group.
  The Trail Making Test (TMT) is widely used in both research and clinical settings as a test of some aspects of executive function. Subtracting TMT A completion time from that of TMT B (TMT B-A) is thought to allow the relative contributions of visual search and psychomotor speed to be parsed from the more complex executive functions (such as cognitive flexibility) required to alternate between numbers and letters. Lower scores indicated better cognitive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Vega, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vega Lab Website — https://www.vegaresearchlab.com